## Suppression of Phoenixin-14 Predicts Mortality in Sepsis: Evidence from Serum Levels and Gene Expression

Assistant Professor, MD Gülsüm ALTUNTAŞ

30.04.2024

Department of Anesthesiology and Reanimation, Firat University Medicine Faculty Hospital, Elazig 23300, Turkey

## INFORMED CONSENT FORM FOR RESEARCH PURPOSES

This study entitled "Investigation of the Correlation Between PNX-14 Levels and Anti-Inflammatory Cytokines and Disease Course in Sepsis Patients in the Intensive Care Unit" aims to identify biomolecules associated with increased inflammation in patients diagnosed with sepsis.

Sepsis is one of the leading causes of critical illness and mortality among patients admitted to the intensive care unit (ICU). It is defined as a life-threatening organ dysfunction caused by a dysregulated host response to infection. In sepsis, the interaction between the causative microorganism and a genetically susceptible host triggers an inflammatory response, resulting in the release of biomarkers that may reflect the severity and progression of the disease. When a microorganism enters the body, the immune system is activated and multiple inflammatory mediators are released. At the same time, the body's defense mechanisms initiate an anti-inflammatory response, leading to the secretion of certain anti-inflammatory substances.

In this study, we aim to compare inflammatory and anti-inflammatory responses in patients diagnosed with sepsis and to investigate the potential protective role of an anti-inflammatory molecule known as Phoenixin-14 in sepsis patients. For this reason, we invite you/your relative who is currently hospitalized in our intensive care unit to participate in this study.

This study is conducted solely for research purposes, and participation is entirely voluntary. The laboratory analyses will be performed using blood samples that are already routinely collected as part of standard intensive care follow-up. From these routinely collected blood samples, 2 mL of blood will be separated for research purposes without affecting routine clinical care. No additional blood samples will be taken, and no extra laboratory tests will be requested.

The study involves the evaluation of daily consciousness level, blood pressure, clinical status, and laboratory parameters of you/your patient. All monitoring and follow-up procedures will be carried out by the physicians and nurses working in the intensive care unit. No additional medical intervention will be performed within the scope of this research, and no tests or procedures outside standard intensive care practice will be requested or applied. Participation in this study does not pose any additional risk or discomfort beyond routine intensive care treatment.

However, since we wish to review certain medical data and laboratory values belonging to you/your patient, this informed consent form has been prepared to obtain your permission. If you consent to the use of this information for scientific purposes, provided that personal identifiers remain confidential, you will be asked to sign this form. All data will be used solely for scientific purposes and handled in accordance with confidentiality and data protection principles.

This research is conducted under the responsibility of Dr. Faculty Member Gülsüm Altuntaş, Department of Anesthesiology and Reanimation.

Statement of the Participant / Patient

| Participant: |
|--------------------------------------------------------------|
| Name and surname: |
| Address: |
| Telephone: |
| Signature: |
| Witness to the interview: |
| Name and surname: |
| Address: |
| Telephone: |
| Signature: |
| Physician conducting the interview: |
| Name, surname, and title: Dr. Faculty Member Gülsüm ALTUNTAŞ |
| Address: Fırat University Faculty of Medicine, |
| Department of Anesthesiology and Reanimation |
| Telephone: +90 541 634 8649 |
| Signature: |